CLINICAL TRIAL: NCT02410460
Title: The Use of Propofol/Ketamine Anesthesia With Bispectral Monitoring (PKA-BIS) Versus Inhalational Anesthetics in Rhytidoplasty - A Prospective, Double-blinded, Randomized Comparison Study
Brief Title: Anesthetics in Rhytidoplasty - A Comparison Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mercy Facial Plastic Surgery Center (Other)
Responsible Party: Principal Investigator, Kristin A. Jones, Principal Investigator, Mercy Facial Plastic Surgery Center
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: MercyFPSC
Record Dates: First submitted 2015-02-23; First posted 2015-04-07 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Rhytidoplasty
MeSH Terms: interventions — Clonidine; Glycopyrrolate; Propofol; Ketamine; Bupivacaine; Scopolamine; Midazolam; Metoclopramide; Lidocaine; Famotidine; Desflurane; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PKA-BIS (intravenous anesthesia) (Other): Received the following medications:
  clonidine 0.1-0.2mg glycopyrrolate 0.2mg propofol infusion titrated to BIS of 60-75 ketamine 50mg + additional ketamine not to exceed 200mg aggregate dosage throughout the case local anesthetic (lidocaine/marcaine mix)
  Interventions: Drug: clonidine; Drug: glycopyrrolate; Drug: propofol; Drug: ketamine; Drug: marcaine; Drug: lidocaine
- Inhalational anesthesia (Other): Received the following:
  Pre-operatively:
  famotidine 20mg scopolamine 1.5mg transdermal patch midazolam 2mg ondansetron 8mg metoclopramide 10mg glycopyrrolate - dose determined by anesthesiologist
  During the case, medication choices and dosing were dependent on the anesthesiologist - all general anesthesia cases received inhalational anesthetic (type of anesthetic - desfluorane vs. sevofluorane - also varied based on anesthesiologist's choice)
  Interventions: Drug: clonidine; Drug: marcaine; Drug: scopolamine; Drug: midazolam; Device: ondansetron; Drug: metoclopramide; Drug: glycopyrrolate; Drug: lidocaine; Drug: famotidine; Drug: desflurane; Drug: sevoflurane

INTERVENTIONS:
Drug: clonidine
Drug: glycopyrrolate
  Arms: PKA-BIS (intravenous anesthesia)
Drug: propofol
  Arms: PKA-BIS (intravenous anesthesia)
Drug: ketamine
  Arms: PKA-BIS (intravenous anesthesia)
Drug: marcaine
Drug: scopolamine
  Arms: Inhalational anesthesia
Drug: midazolam
  Arms: Inhalational anesthesia
Device: ondansetron
  Arms: Inhalational anesthesia
Drug: metoclopramide
  Arms: Inhalational anesthesia
Drug: glycopyrrolate
  Arms: Inhalational anesthesia
Drug: lidocaine
Drug: famotidine
  Arms: Inhalational anesthesia
Drug: desflurane
  Arms: Inhalational anesthesia
Drug: sevoflurane
  Arms: Inhalational anesthesia

SUMMARY:
This study is a prospective, double-blind, randomized comparison study of different anesthesia methods in rhytidoplasty surgery. The study is designed to determine whether post-operative side-effect profiles in patients undergoing elective cosmetic facelift surgery can be decreased through the use of propofol/ketamine anesthesia with bispectral monitoring (PKA-BIS) rather than general anesthesia, without increasing intra-operative time, side-effect profiles, or patient recall. Approximately 30 subjects undergoing facelift surgery performed by the principal investigator will participate.

DETAILED DESCRIPTION:
PKA-BIS arm receives the following medications:

clonidine 0.1-0.2mg glycopyrrolate 0.2mg propofol infusion titrated to BIS of 60-75 ketamine 50mg + additional ketamine not to exceed 200mg aggregate dosage throughout the case local anesthetic (lidocaine/marcaine mix)

General Anesthesia arm receives the following medications:

Pre-operatively:

Pepcid 20mg Scopolamine 1.5mg transdermal patch Versed 2mg Zofran 8mg Reglan 10mg Glycopyrrolate - dose determined by anesthesiologist

During the case, medication choices and dosing were dependent on the anesthesiologist - all general anesthesia cases received inhalational anesthetic (type of anesthetic also varied based on anesthesiologist's choice)

ELIGIBILITY:
Inclusion criteria:

* Female
* 18 years of age or older
* Undergoing elective rhytidoplasty

Exclusion criteria:

* Male
* Under 18 years old
* Pregnant or breastfeeding
* Medically unfit to undergo surgery
* Undergoing brow-lift in conjunction with rhytidoplasty (due to the inability to properly secure the BIS monitor as it would lie within the surgical field)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Pain (QOR-40/VAS) | 1 week
  Quality of recovery score (QOR-40) in PACU and POD#1, VAS POD#1 and POD#7
Nausea/vomiting (QOR-40) | 24 hours
  Quality of recovery score (QOR-40) in PACU and POD#1
Time to awakening | 4 hours
  staff recorded
Time to discharge | 4 hours
  staff recorded
Overall feeling of well-being (QOR-40/VAS) | 1 week
  Quality of recovery score (QOR-40) in PACU and POD#1, VAS POD#1 and POD#7

SECONDARY OUTCOMES:
Cost (reported as a mean) | 1 day
  comparison between two groups (reported as a mean)

CONTACTS AND LOCATIONS:
Locations (1):
- Mercy Facial Plastic Surgery Center, Springfield, Missouri, United States

REFERENCES:
- [Derived] Jones KA, LaFerriere KA. Intravenous Anesthesia With Bispectral Index Monitoring vs Inhalational Anesthesia for Rhytidoplasty: A Randomized Clinical Trial. JAMA Facial Plast Surg. 2015 Jul-Aug;17(4):239-44. doi: 10.1001/jamafacial.2015.0222. PMID 25906190